CLINICAL TRIAL: NCT07254715
Title: Does Itopride Improve Semaglutide Induced Gastroparesis Ultrasound Before Anesthesia? Randomized Controlled Trial
Brief Title: Effect of Itopride on Semaglutide Gastroparesis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Tamer Samir Abdelsalam, Assistant professor of anesthesia, Intensive care and Pain medicine, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FMASU R263/2025
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Semaglutide-Induced Gastric Motility; Anesthesia
Keywords: itopride; gastric ultrasound

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Itopride HCL (Active Comparator): Daily oral 50mg Itopride tablet TID, 1 hour before meals for 7 days
  Interventions: Drug: Itopride HCI 50 mg
- Placebo (Placebo Comparator): Daily placebo tablet TID, 1 hour before meals for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Itopride HCI 50 mg — Daily oral 50mg Itopride tablet TID, 1 hour before meals for 7 days
  Arms: Itopride HCL
Drug: Placebo — Daily placebo tablet TID, 1 hour before meals for 7 days
  Arms: Placebo

SUMMARY:
Semaglutide delays gastric emptying and increases the risk of aspiration with anesthesia; So, the addition of prokinetics as Itopride, could enhance gastric emptying and hasten surgery.

The investigator will evaluate the effect of Itopride on Semaglutide-induced gastroparesis and residual gastric contents after 8 hours of fasting by gastric ultrasound before anesthesia.

DETAILED DESCRIPTION:
Semaglutide delays gastric emptying and increases the risk of aspiration with anesthesia; So, the addition of prokinetics as Itopride could enhance gastric emptying and hastens surgery.

Semaglutide, a glucagon-like peptide-1 (GLP-1) agonist, is gaining popularity for the treatment of type 2 diabetes mellitus (T2DM) and obesity; Semaglutide stimulates insulin excretion and delays gastric emptying.Itopride, a novel prokinetic agent, acts as a dopamine D2 receptor antagonist and an acetylcholine esterase inhibitor. Itopride shows promise in managing gastroparesis symptoms by accelerating gastric emptying, improving gastric tension and sensitivity, and exerting antiemetic effects.

The investigator designed this prospective, randomized, double-blind controlled study to evaluate the effect of Itopride on Semaglutide induced gastroparesis and residual gastric contents after 8-hours fasting by gastric ultrasound before anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists grade I- III.
* Age: 40-60 years.
* BMI: 20-30 kg/m2.
* Diabetic patients on semaglutide (0.5-1mg) SC weekly.
* Undergoing elective hysterectomy.

Exclusion Criteria:

* Declining to give written informed consent.
* history of upper abdominal surgery or the presence of hiatal hernia.
* Other medications inducing gastroparesis (opioids, proton pump inhibitors, tricyclic antidepressants, calcium channel blockers, antipsychotic medications, and lithium).
* History of allergy to Itopride.
* History of cardiac arrhythmia or abnormal ECG.
* Neurologic diseases (including Parkinson's disease and multiple sclerosis)
* Hepatic or renal failure.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Residual gastric contents | on day 7
  Residual gastric contents (clear fluid ˃1.5 mL/kg or the presence of solids) by ultrasound in the right lateral decubitus after 8-hours fasting .

SECONDARY OUTCOMES:
Residual gastric contents on day 3 and day 5. | on day 3 and day 5
Incidence of vomiting during anesthesia | during anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of medicine, Ain Shams University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No